CLINICAL TRIAL: NCT05863923
Title: mHealth Messaging to Motivate Quitline Use and Quitting Among Persons Living With HIV (PLWH) in Vietnam (M2Q2-HIV)
Brief Title: Tobacco Cessation Texting Intervention for People Living With HIV Who Smoke in Vietnam
Acronym: M2Q2-HIV
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Institute of Population, Health and Development, Vietnam (Other)
Responsible Party: Principal Investigator, Rajani Sadasivam, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H00023608; U01CA261604 (NIH)
Record Dates: First submitted 2023-03-31; First posted 2023-05-18 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Tobacco Cessation
Keywords: mHealth
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Seroconversion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The M2Q2-HIV intervention includes 3 functions: 1) Extended CHW services, 2) M2Q2 computer-tailored peer messaging, and 3) texting facilitation to quitline use and the quitline intervention. Our goals are to promote the use of an underused, available, government-funded resource for public health (quitline) and NRT that the quitline provides, thus promoting smoking cessation among PLWH.
  Interventions: Behavioral: mHealth Messaging to Motivate Quitline use and Quitting among Persons Living With HIV (PLWH) in Vietnam (M2Q2-HIV)
- Comparison (Active Comparator): Comparison smokers will receive five brief "risk of smoking" texts as minimal texting intervention, to enhance blinding to knowledge of randomization group.
  Interventions: Behavioral: M2Q2-HIV Comparison

INTERVENTIONS:
Behavioral: mHealth Messaging to Motivate Quitline use and Quitting among Persons Living With HIV (PLWH) in Vietnam (M2Q2-HIV) — Participants in the intervention group will be exposed to the texting intervention through a series of culturally tailored assessments and motivational text messages from the text messaging system sent throughout the 6 months of duration of the study.
  Arms: Intervention
Behavioral: M2Q2-HIV Comparison — Participants in the comparison group will be exposed to a brief set of five texts with facts about smoking risks and assessment messages that are not culturally tailored from the text messaging system.
  Arms: Comparison

SUMMARY:
The intersection of smoking and HIV/AIDS poses a serious public health threat in Vietnam. Vietnam is dealing with these two challenges with parallel rather than integrated plans. Using a computer-tailored texting intervention, study investigators seek to promote the use of an underused, available, government-funded resource (the Quitline) and Nicotine Replacement Therapy (NRT) that the quitline provides, thus, promoting cessation among PLWH.

DETAILED DESCRIPTION:
M2Q2-HIV [mHealth Messaging to Motivate Quitline Use and Quitting among Persons Living with HIV (PLWH) in Vietnam (M2Q2-HIV)] is an adaptation of a current computer-tailored smoking cessation intervention in Vietnam. Study investigators seek to promote underused government resources for public health (the Quitline) and Nicotine Replacement Therapy (NRT) among PLWH in a sustainable manner.

Investigators will test M2Q2-HIV by conducting a randomized control trial with 600 PLWH smokers in two provinces in Northern Vietnam (26 clinics; 9,877 HIV patients).

In Aim 1, study investigators will conduct formative work to prepare the M2Q2-HIV system for PLWH smokers.

In Aim 2, the study team will randomize and follow smokers for six months. The study's effectiveness hypothesis will evaluate carbon monoxide (CO) verified, six-month, seven-day point prevalence cessation. Process hypotheses will evaluate self-efficacy, Quitline, and NRT use and test our hypothesized model that specific measured processes will partially mediate observed intervention effectiveness.

Using qualitative interviews with key stakeholders and PLWH smokers, Aim 3 will support nationwide M2Q2-HIV dissemination assessing acceptability and contextual factors guided by the Practical, Robust Implementation and Sustainability Model (PRISM).

This project builds upon a long-standing, successful collaboration between institutions in Vietnam (Ministry of Health, Bach Mai Quitline, Institute of Population Health and Development, Hanoi Medical University) and UMass Chan Medical School. The study team has expertise in smoking cessation, HIV intervention, including stigma related to concomitant substance use, and implementation of complex interventions. If proven effective, the Vietnam Ministry of Health is committed to incorporating M2Q2-HIV as a permanent part of the national infrastructure.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed HIV infection (prevalent and incident HIV).
2. At least 18 years old.
3. Current smoker.
4. Be able to receive texts and read text (literate).

Exclusion Criteria:

1. Pregnant or planning to become pregnant during the next six months.
2. Unable or unwilling to provide informed consent.
3. Prior diagnosis of serious mental health illness.
4. Smoker who helped develop the motivational texts used in the intervention (participated in Aim 1).
5. Family member of another participant in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Smoking Cessation Rate | At 6 months post-randomization
  At six months, we will assess 7-day point prevalence cessation, based on the following question: "Do you currently smoke tobacco (smoked even 1 puff in the last 7 days)?" The Society of Nicotine and Tobacco Research has recommended this measure.

SECONDARY OUTCOMES:
Self-Efficacy | 0-month (baseline) and 6-months post-randomization
  Self-Efficacy, as measured by the Smoking Self-Efficacy Questionnaire (SEQ-12) questionnaire. The score for each question ranges on a 4-point Likert scale from 0-3. SEQ-12 score ranges from 0-36, with higher values indicating higher self-efficacy for smoking cessation. The aggregate score will only be computed if no more than 2 out of the 12 questionnaire items had missing or 'not applicable' responses.
HIV-Related Stigma | 0-month (baseline) and 6-months post-randomization
  HIV-related stigma, measured using a survey assessing five indicators of HIV/AIDS-related stigma according to USAID: (1) blame, judgment; (2) shame; (3) enacted stigma/discrimination; (4) disclosure; and (5) fear of casual transmission and refusal of contact. Survey response options include (1) Yes, (2) No, and (3) No answer. A response of "yes" to one or more survey questions will indicate the presence of HIV-related stigma.
Quitline Use | 6-months post-randomization
  The quitline staff will record details of intake assessment (time on call, readiness to quit, quit date, and goal-setting) and fidelity of follow-up call completion.
NRT Use | 6-months post-randomization
  The quitline staff will document the distribution of NRT lozenge and smoker use of NRT during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rajani S Sadasivam, PhD, Principal Investigator — University of Massachusetts Chan Medical School; Hoa T Nguyen, MD, MS, PhD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (2):
- UMass Chan Medical School, Worcester, Massachusetts, United States
- Institute of Population, Health, and Development (PHAD), Hanoi, Vietnam